CLINICAL TRIAL: NCT00216463
Title: A Phase 2, Randomized, Double Blind, Placebo-Controlled, Parallel Group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Varying Loading and Maintenance Dosing Regimens of ISIS 301012 Administered to Hypercholesterolemic Subjects
Brief Title: Safety and Tolerability of Varying Load and Dose of ISIS 301012 in People With Elevated LDL-cholesterol Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Medical Monitor, Genzyme Coporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 301012CS3; EudraCT No.: 2004-003934-32
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Hypercholesterolemia
Keywords: LDL-cholesterol; apoB-100; apoB-48
MeSH Terms: conditions — Hypercholesterolemia | interventions — mipomersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- A (Experimental): Slow load with every other week maintenance
  Interventions: Drug: ISIS 301012 or Placebo
- B (Experimental): Slow load with every other week maintenance
  Interventions: Drug: ISIS 301012 or Placebo
- C (Experimental): No load; once weekly maintenance
  Interventions: Drug: ISIS 301012 or Placebo
- D (Experimental): No load; once weekly maintenance
  Interventions: Drug: ISIS 301012 or Placebo
- E (Experimental): No load; once weekly maintenance
  Interventions: Drug: ISIS 301012 or Placebo

INTERVENTIONS:
Drug: ISIS 301012 or Placebo — 200 mg subcutaneous injection - 4 loading doses within the first 11 days followed by: 200 mg subcutaneous injection - every other week for 11 weeks
  Arms: A
Drug: ISIS 301012 or Placebo — 200 mg subcutaneous injection - 4 loading doses within the first 11 days followed by: 100 mg subcutaneous injection - every other week for 11 weeks
  Arms: B
Drug: ISIS 301012 or Placebo — 300 mg subcutaneous injection - every week for 13 weeks
  Arms: D
Drug: ISIS 301012 or Placebo — 400 mg subcutaneous injection - every week for 13 weeks
  Arms: E
Drug: ISIS 301012 or Placebo — 200 mg subcutaneous injection - every week for 13 weeks
  Arms: C

SUMMARY:
The aim of this study is to assess the safety and tolerability of varying dose and load regimens of ISIS 301012 in people who have elevated LDL-cholesterol levels.

ELIGIBILITY:
Inclusion Criteria:

* BMI >/= 25 to </= 32 kg/m^2
* fasting stable LDL-cholesterol >/= 130 mg/dL (3.36 mmol/L) and triglycerides < 400 mg/dL (4.55 mmol/L)
* Females not of childbearing potential

Exclusion Criteria:

* No endocrine, hematologic, renal, hepatic, metabolic, psychiatric, neurology, pulmonary or cardiovascular disease
* Subjects who test positive for hepatitis B, C or HIV
* Current diagnosis or known history of liver disease, such as acute or chronic hepatitis, liver cirrhosis, liver steatosis, or liver function abnormalities such as AST, ALT, GGT, or total bilirubin >/= 1.5 x ULN at Screening
* A systolic blood pressure >/= 160 mmHg or a diastolic blood pressure >/= 95 mmHg on 2 occasions during Screening
* Concomitant medications within 14 days of dosing, except hormone replacement therapy for post-menopausal women and acetylsalicylic acid or paracetamol dosed for fewer than five consecutive days
* Subject has taken any lipid-lowering drug within 30 days or five half-lives (of the lipid-lowering drug) whichever is longer, prior to Screening
* Alcohol or drug abuse within 2 years of Screening
* Donated blood (450 mL) within the 3 months prior to Screening or suffered significant blood loss equal to a blood donor portion
* Subject smokes > 10 cigarettes, or more than one pipe or one cigar per day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-08; Primary Completion 2007-03 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Percent reduction in LDL-cholesterol from baseline | 14 days post dosing

SECONDARY OUTCOMES:
Percent reduction in apoB-100 from baseline | 14 days post dosing
Percent change from baseline in HDL-cholesterol, triglycerides, total cholesterol, non-HDL cholesterol, VLDL and LP(a) | 14 days post dosing
Percent change from baseline in LDL/HDL and apoB-100/apo-A1 ratios | 14 days post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Berlin, Germany

REFERENCES:
- [Derived] Akdim F, Tribble DL, Flaim JD, Yu R, Su J, Geary RS, Baker BF, Fuhr R, Wedel MK, Kastelein JJ. Efficacy of apolipoprotein B synthesis inhibition in subjects with mild-to-moderate hyperlipidaemia. Eur Heart J. 2011 Nov;32(21):2650-9. doi: 10.1093/eurheartj/ehr148. Epub 2011 May 18. PMID 21593041